CLINICAL TRIAL: NCT06589102
Title: Prevalence and Consequences of Hyperlactemia Following Pancreatic Surgery
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Grip, Primary investigator, Karolinska University Hospital
Other Study IDs: 2019-04284
Record Dates: First submitted 2023-05-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer; Pancreatic Cyst; Chronic Pancreatitis
Keywords: Pancreatic surgery
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate the role of lactate elevation.

The main aims are:

* Determine the frequency of lactate elevation following pancreatic surgery and its relationship to postoperative complications
* Investigate what patient and surgical related factors that are associated with postoperative lactate elevation This is a retrospective study based on existing medical data and will not affect the medical care of the studied patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreatic surgery 2016-2018

Exclusion Criteria:

* Patients unable to undergo scheduled surgery
* Missing data in the postoperative period

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients scheduled to undergo major pancreatic surgery in a tertiary university hospital during 2016-18
Sampling Method: Non-Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | All patients are followed until they leave the hospital, but a maximum of six months
  hospital stay following surgery

SECONDARY OUTCOMES:
General postoperative complications | All patients are followed until they leave the hospital, but a maximum of six months
  Defined as Clavien-Dindo grade III-V
ICU care | All patients are followed until they leave the hospital, but a maximum of six months
  Organ failure requiring ICU care
Surgery specific complications | 90 days
  Pancreatic fistula, bile leakage, delayed gastric emptying

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden